CLINICAL TRIAL: NCT01522508
Title: Detection of Nociceptive Stimulation by Analgesia Nociception Index (ANI) During Anesthesia With Propofol or Sevoflurane and Varying Remifentanil Concentrations.
Brief Title: Evaluation of Analgesia Nociception Index (ANI) During Propofol/Remifentanil and Sevoflurane/Remifentanil Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Berthold Bein, Prof. Dr. med., University Hospital Schleswig-Holstein
Other Study IDs: ANI-134-1
Record Dates: First submitted 2012-01-26; First posted 2012-01-31 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: General Anaesthesia
Keywords: Analgesia; Anesthetics; Diagnostic Techniques and Procedures
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- propofol/remifentanil: patients receive standardized propofol and changing remifentanil concentrations
  Interventions: Procedure: tetanic stimulation
- sevoflurane/remifentanil: patients receive standardized sevoflurane and changing remifentanil concentrations
  Interventions: Procedure: tetanic stimulation

INTERVENTIONS:
Procedure: tetanic stimulation — as test stimulus a painful tetanic stimulation is used

SUMMARY:
The aim of this prospective randomized study was to evaluate the ability of the new Analgesia Nociception Index ANI, derived by heart rate variability, to detect painful stimulation during either propofol or sevoflurane anesthesia and changing remifentanil concentrations.

DETAILED DESCRIPTION:
Monitoring Antinociception during general anesthesia is still a big challenge in the field and has not become clinical routine yet. Recently, for the Surgical Pleth Index SPI a benefit for the patient in terms of reduction of remifentanil use, less unwanted effects and shorter recovery from anesthesia was reported. However, there are new variables like the ANI that are developed to measure antinociception during anesthesia.

In the present study the investigators want to evaluate, whether ANI detects a painful tetanic stimulus during general anesthesia using propofol or sevoflurane and different concentrations of remifentanil.

ELIGIBILITY:
Inclusion Criteria:

* age between 18- 65 years,
* ASA physical status I or II,
* elective surgery in general anesthesia planned,
* written informed consent

Exclusion Criteria:

* pregnancy,
* history of cardiac arrhythmia,
* presents of any neuromuscular or neurologic disease,
* use of CNS-active medication or abuse of alcohol/illicit drugs -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery in general anesthesia
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-07 (Estimated); Study Completion 2012-10 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Kiel, Dept. of Anesthesiology and Intensive Care Med., Kiel, Germany

REFERENCES:
- [Background] Gruenewald M, Meybohm P, Ilies C, Hocker J, Hanss R, Scholz J, Bein B. Influence of different remifentanil concentrations on the performance of the surgical stress index to detect a standardized painful stimulus during sevoflurane anaesthesia. Br J Anaesth. 2009 Oct;103(4):586-93. doi: 10.1093/bja/aep206. Epub 2009 Jul 31. PMID 19648155
- [Background] Struys MM, Vanpeteghem C, Huiku M, Uutela K, Blyaert NB, Mortier EP. Changes in a surgical stress index in response to standardized pain stimuli during propofol-remifentanil infusion. Br J Anaesth. 2007 Sep;99(3):359-67. doi: 10.1093/bja/aem173. Epub 2007 Jul 3. PMID 17609248
- [Derived] Gruenewald M, Ilies C, Herz J, Schoenherr T, Fudickar A, Hocker J, Bein B. Influence of nociceptive stimulation on analgesia nociception index (ANI) during propofol-remifentanil anaesthesia. Br J Anaesth. 2013 Jun;110(6):1024-30. doi: 10.1093/bja/aet019. Epub 2013 Mar 6. PMID 23471754